CLINICAL TRIAL: NCT00661726
Title: A Phase IIA Study of Subcutaneous 5-aza-2'- Deoxycytidine (Decitabine) in Patients With Thalassemia Intermedia
Brief Title: Evaluating the Safety and Effectiveness of Decitabine in People With Thalassemia Intermedia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 569; U01HL065238 (NIH); 68,995
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-02

CONDITIONS: Thalassemia
Keywords: Thalassemia Intermedia
MeSH Terms: conditions — Thalassemia; beta-Thalassemia | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will receive injected decitabine for 12 weeks.
  Interventions: Drug: Decitabine (USAN, INN)

INTERVENTIONS:
Drug: Decitabine (USAN, INN) — Participants will receive 0.2 mg/kg of decitabine subcutaneously twice a week for 12 weeks. The dose will be reduced for toxicities as needed. The maximum dose of decitabine to be given will be 0.2 mg/kg.
  Other Names: 5-aza-2'-deoxycytidine (NCS 127716); DAC; 5-Aza-CdR; Deoxyazacytidine; 1-(2'deoxy-D-ribofuranosy1)-5-azacytosine; Dezocitidine; Dacogen

SUMMARY:
Thalassemia intermedia (TI) is an inherited blood disorder that can cause anemia due to low levels of hemoglobin. Decitabine is a medication that may be effective at increasing hemoglobin levels. This study will evaluate the safety and effectiveness of decitabine at increasing hemoglobin levels in people with TI.

DETAILED DESCRIPTION:
Thalassemias are inherited blood disorders that are characterized by low levels of hemoglobin and healthy red blood cells, which can lead to anemia. There are many different types of thalassemias, and TI is one type. People with TI often have moderate to severe anemia and may have a shortened life span, organ damage, and a lower quality of life as a result of the disease. Decitabine is a medication used to treat people with diseases that affect bone marrow and blood cells. The medication may be an effective treatment for people with TI because it may have the ability to interact with a person's DNA and increase hemoglobin levels. Previous studies in people with anemia have shown that decitabine has increased hemoglobin levels in some participants. The purpose of this study is to evaluate the safety and effectiveness of decitabine at increasing hemoglobin levels in people with TI.

This study will enroll people with TI. Following an 8-week screening period, participants will attend a baseline study visit, which will include a blood collection, pregnancy test, physical exam, and echocardiogram heart imaging procedure. Decitabine will be injected under the skin in the abdomen, thigh, or upper arm. Participants will be observed for a minimum of 30 minutes after the injection to assess pain or adverse reactions. Participants will then receive low doses of decitabine twice a week, on consecutive days, for 12 weeks. They will be closely monitored and dosages will be adjusted or stopped as needed. Every 2 weeks, participants will undergo a blood collection for safety testing. Every 4 weeks, participants will attend a study visit for a pregnancy test, physical exam, blood collection, and review of medication effects. Additionally, at the Week 12 visit, a repeat echocardiogram will occur. During Weeks 12 to 24, participants will not receive decitabine injections but will attend monthly study visits for repeat testing. Study researchers will contact participants by phone every 3 months during Year 1 and then every 6 months for the duration of the study to collect long-term survival and medical information.

ELIGIBILITY:
Inclusion Criteria:

* Beta-thalassemia and beta thalassemia-hemoglobin E (HbE), as confirmed by DNA testing
* Transfusion independent for at least 120 days before study entry
* Red blood cell folate levels above the lower limit of normal

Exclusion Criteria:

* Absolute neutrophil count (ANC) less than 2000/mm3 in the 8 weeks before study entry or a history of chronic neutropenia, defined as an ANC less than 2000/mm3
* Platelet count less than 100,000/mm3 or greater than 1,000,000/mm3 in the 8 weeks before study entry
* Family history of an inherited disease resulting in low ANC or bone marrow failure
* Serum creatinine level greater than 2 mg/dL in the 8 weeks before study entry
* Evidence of liver disease, as defined by one or more of the following conditions:

  1. Alanine aminotransferase (ALT) level greater than 3 times the upper limit of normal in the 8 weeks before study entry
  2. Serum albumin level less than 3 g/dL in the 8 weeks before study entry
  3. Evidence of cirrhosis on liver biopsy obtained in the 6 months before study entry
* Approaching death; has concurrent liver, kidney, cardiac, or metabolic disease; or has any disease of such severity that death within 7 to 10 days of study entry is likely
* Pregnant, planning to become pregnant, or breastfeeding
* Sexually active female of childbearing potential who is unwilling to use at least two acceptable methods of contraception, as determined by the investigator
* Sexually active male whose partner is of child-bearing potential and who is unwilling to use at least two acceptable methods of contraception, as determined by the investigator, during and for 2 months after decitabine treatment
* Diagnosed with cancer (except non-melanoma skin cancer) in the 5 years before study entry. In particular, suspicion or evidence of myelodysplastic syndrome (MDS) on clinically indicated bone marrow aspirate or a family history of MDS or concurrent leukemia
* HIV infection
* Not expected to be able to complete 24 weeks of study follow-up
* Currently being treated with any experimental or fetal hemoglobin modulating agent
* Current participation in any other studies of investigational drugs or devices
* Unable to comply with study medication regimen
* Any condition, which in the opinion of the investigator, would place the individual at undue risk if treated with twice-weekly low-dose decitabine for 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Olivieri, MD, Study Chair — University Health Network/Toronto General Hospital
Locations (3):
- United States (2):
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital Philadelphia, Philadelphia, Pennsylvania
- University Health Network, Toronto, Canada

REFERENCES:
- [Result] Olivieri NF, Saunthararajah Y, Thayalasuthan V, Kwiatkowski J, Ware RE, Kuypers FA, Kim HY, Trachtenberg FL, Vichinsky EP; Thalassemia Clinical Research Network. A pilot study of subcutaneous decitabine in beta-thalassemia intermedia. Blood. 2011 Sep 8;118(10):2708-11. doi: 10.1182/blood-2011-03-341909. Epub 2011 Jun 23. PMID 21700776

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in early 2007 at one site, Toronto General Hospital. When recruitment became too challenging, the study was moved to the Thalassemia Clinical Research Network and opened at 2 more sites in 2008. These included Children's Hospital in Philadelphia and Children's Hospital in Oakland. Recruitment closed in May, 2010 with 6 subjects.
Pre-assignment Details: To be eligible, patients had to be >=18 years of age and have beta thalassemia intermedia or beta thalassemia-HbE intermedia, no transfusions for 120 days, no hydroxyurea for 120 days, have RBC folate levels above the lower limit of normal, and steady-state anemia (post pt #2, the protocol was amended to define anemia hemoglobin level of <10g/dl).
Groups:
- Phase IIA Open Label, Single-arm, Multi-center Pilot Study: Participants will receive injected decitabine for 12 weeks.
Period: Overall Study
Arm/Group | Phase IIA Open Label, Single-arm, Multi-center Pilot Study
Started | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Phase IIA Open Label, Single-arm, Multi-center Pilot Study
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 3
  Canada | 3
Patients that had been splenectomized [Number; unit: participants]
  Yes | 5
  No | 1
Received transfusion in preceding year but > 120 days before protocol therapy [Number; unit: participants]
  Yes | 4
  No | 2
Baseline Hemoglobin [Mean (Standard Deviation); unit: g/dl] | 7.9 (1.8)
Documented Concomitant Mutation at the alpha-globin locus [Number; unit: participants]
  Yes | 1
  No | 5

OUTCOME MEASURES:

1. Secondary Outcome: Change in Absolute Fetal Hemoglobin (HbF) From Baseline to Peak (the Follow-up Time Point With the Highest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: g/dL
Groups:
- Decitabine: Decitabine 0.2 mg/kg was administered subcutaneously daily on the same 2 consecutive days each week for 12 weeks.
Arm/Group | Decitabine
Number analyzed (Participants) | 5
g/dL | 0.65 (0.06)
Statistical Analysis 1: Comparison: Decitabine; Linear regression after adjusting for time duration was used to test the mean difference between baseline and follow-up values; Test type: Superiority or Other; p < 0.01, Regression, Linear

2. Primary Outcome: Number of Evaluable Patients With an Increase From Baseline in Hemoglobin (Hb) of ≥1.5 g/dL
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Number; unit: participants
Arm/Group | Decitabine
Number analyzed (Participants) | 5
participants | 2

3. Secondary Outcome: Change in Indirect Bilirubin From Baseline to Nadir (the Follow-up Time Point With the Lowest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Decitabine
Number analyzed (Participants) | 5
µmol/L | -17.36 (6.95)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.045, Regression, Linear

4. Secondary Outcome: Change in Serum Lactate Dehydrogenase (LDH) From Baseline to Nadir (the Follow-up Time Point With the Lowest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Decitabine
Number analyzed (Participants) | 5
U/L | -116.60 (40.81)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.083, Regression, Linear

5. Secondary Outcome: Change in Absolute Reticulocyte Count From Baseline to Nadir (the Follow-up Time Point With the Lowest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: X (10^9)/L
Arm/Group | Decitabine
Number analyzed (Participants) | 5
X (10^9)/L | -34.00 (12.50)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.039, Regression, Linear

6. Secondary Outcome: Change in Erythropoietin Levels From Baseline to Nadir (the Follow-up Time Point With the Lowest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: mIU/mL
Arm/Group | Decitabine
Number analyzed (Participants) | 5
mIU/mL | -43.78 (21.60)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.18, Regression, Linear

7. Secondary Outcome: Change in Platelet Count From Baseline to Peak (the Follow-up Time Point With the Highest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: X (10^9)/L
Arm/Group | Decitabine
Number analyzed (Participants) | 5
X (10^9)/L | 355.0 (102.0)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Regression, Linear

8. Secondary Outcome: Change in Neutrophil Counts From Baseline to Nadir (the Follow-up Time Point With the Lowest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: X (10^9)/L
Arm/Group | Decitabine
Number analyzed (Participants) | 5
X (10^9)/L | -3.15 (1.03)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.069, Regression, Linear

9. Secondary Outcome: Change in Red Blood Cell (RBC) Deformability From Baseline to Peak (the Follow-up Time Point With the Highest Value)
Description: Deformability was assessed by ektacytometry. Normal RBC have maximal deformability, measurable by osmotic ektacytometry, at isotonicity (290 mosmol). A decrease on the Deformability Index (measured in arbitrary units) corresponds to an impairment in the cell membrane's ability to alter its shape under stress.
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: Arbitrary Units
Arm/Group | Decitabine
Number analyzed (Participants) | 5
Arbitrary Units
  Baseline | 0.43 (0.03)
  Change From Baseline | 0.09 (0.05)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.18, Regression, Linear

10. Secondary Outcome: Change in Percentage of Red Blood Cell (RBC) Hb Concentration From Baseline to Peak (the Follow-up Time Point With the Highest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: % of RBC Hb Concentration
Arm/Group | Decitabine
Number analyzed (Participants) | 5
% of RBC Hb Concentration | 7.06 (1.56)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.022, Regression, Linear

11. Secondary Outcome: Change in Percentage of Annexin-positive Cells From Baseline to Nadir (the Follow-up Time Point With the Lowest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: % of Annexin-Positive Cells
Arm/Group | Decitabine
Number analyzed (Participants) | 5
% of Annexin-Positive Cells | -1.26 (0.55)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.11, Regression, Linear

12. Primary Outcome: Change in Total Hemoglobin (Hb) From Baseline to Peak (the Follow-up Time Point With the Highest Value)
Time Frame: up to 12 weeks
Population: One of 6 enrolled patients withdrew from study after week 2 and was not used for analysis.
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Decitabine
Number analyzed (Participants) | 5
g/dL | 1.16 (0.20)
Statistical Analysis 1: Comparison: Decitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Regression, Linear

ADVERSE EVENTS:
Arm/Group | Decitabine
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=5)
High Platelets Count (Blood and lymphatic system disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=5)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Ocular/ visual- other: Conjunctival Infection (Vascular disorders) | 1 (1)
Radiating Pain in Right Shoulder (General disorders) | 1 (1)
Pain - joint (General disorders) | 1 (1)
Palpitation (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No